CLINICAL TRIAL: NCT04958629
Title: A Prospective Cohort Study on Familial Hypercholesterolemia in Health Examination Population
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2021098
Record Dates: First submitted 2021-06-27; First posted 2021-07-12 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-06

CONDITIONS: Familial Hypercholesterolemia
Keywords: familial hypercholesterolemia; prognosis
MeSH Terms: conditions — Hyperlipoproteinemia Type II | interventions — Receptors, LDL

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- non-FH Group
- FH Group
  Interventions: Other: familial hypercholesterolemia

INTERVENTIONS:
Other: familial hypercholesterolemia — Among the selected patients with hyperlipidemia, those who met the diagnostic criteria of FH were included in the study cohort as FH group.
  Groups: FH Group

SUMMARY:
To determine the prevalence and the prognosis in a corhort of patients with familial hypercholesterolemia (FH).

DETAILED DESCRIPTION:
This study aims to achieve the following goals through prospective cohort study and statistical analysis: (1) to determine the prevalence of familial hypercholesterolemia (FH) in healthy people with hypercholesterolemia.（2) Compared with non FH population, the relative risk of atherosclerotic cardiovascular disease (ASCVD) in FH patients in China was calculated, and the risk prediction model of ASCVD in FH patients was constructed by using biochemical results, imaging data, biomarkers and other indicators.（3) To evaluate the benefits of different lipid-lowering strategies for FH patients in China.（4) To analyze the gene carriers of FH patients in China.

ELIGIBILITY:
Inclusion Criteria:

1) Patients with definite diagnosis of hyperlipidemia.

Exclusion Criteria:

1. Age < 18.
2. Do not agree to participate in this study.
3. secondary hypercholesterolemia.
4. Phytosteronemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hyperlipidemia were screened from health examination population. Among the selected patients with hyperlipidemia, those who met the following inclusion and exclusion criteria were included in the study cohort as FH group or non-FH group.
Sampling Method: Non-Probability Sample
Enrollment: 318 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with atherosclerotic cardiovascular disease (ASCVD) events | 2 years from enrollmet
  1) Fatal or non-fatal myocardial infarction; 2) Fatal or non-fatal ischemic stroke; 3) Coronary artery revascularization; 4) Peripheral artery revascularization; 5) Cardiogenic death

CONTACTS AND LOCATIONS:
Overall Officials: Wei Gao, Doctor, Study Chair — Peking University Third Hospital

IPD SHARING:
Plan to Share IPD: No